CLINICAL TRIAL: NCT02497495
Title: Effects Post-exercise of Biological, Clinical and Metabolic Variables as From Different Temperatures and Times of Immersion Cold Water Application in Active Individuals
Brief Title: Behaviour After Exercise of Biological, Clinical and Metabolic Variables as From Different Temperatures and Times of Immersion Cold Water Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, PhD, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 736.438
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Cryotherapy Effect
Keywords: Immersion; Recovery of Function; Lactate; Creatine Kinase; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- GC (No Intervention): Control group - CG (n = 21), which suffered no recuperative technique
- G1 (Experimental): G1 (n = 21) was subjected to a recovery procedure by immersion cold water for 5 minutes as from 9±1 degrees Celsius
  Interventions: Other: immersion cold water
- G2 (Experimental): G2 (n = 21) was subjected to a recovery procedure by immersion cold water for 5 minutes as from 14±1 degrees Celsius
  Interventions: Other: immersion cold water
- G3 (Experimental): G3 (n = 21) was subjected to a recovery procedure by immersion cold water for 15 minutes as from 9±1 degrees Celsius
  Interventions: Other: immersion cold water
- G4 (Experimental): G4 (n = 21) was subjected to a recovery procedure by immersion cold water for 15 minutes as from 14±1 degrees Celsius
  Interventions: Other: immersion cold water

INTERVENTIONS:
Other: immersion cold water — immersion cold water at different temperatures and exposure times
  Arms: G1; G2; G3; G4

SUMMARY:
Introduction: immersion cold water is a recuperative strategy commonly used, however, are not yet fully understood the real effects of this technique on specific conditions. Objective: To analyze and to compare the effects of the immersion cold water during the intense post-exercise recovery, using different times and temperatures on biological, clinical and metabolic variables. Method: 105 male subjects were divided into five groups: one control group (CG) and four recoveries (G1: 5' at 9±1 degrees Celsius; G2: 5' at 14±1 degrees Celsius; G3: 15' at 9±1 degrees Celsius; G4: 15' at 14±1 degrees Celsius). The volunteers were submitted an exhaustion protocol that consisted of a program of jumps and the Wingate test. Immediately after the exhaustion protocol, volunteers were directed to a tank with water and ice, which were immersed up to the height of the anterior superior iliac spine to the recovery procedure, during which blood samples were collected for later analysis lactate and creatine kinase (CK). Variables were collected prior to the exercise, 24, 48, 72 and 96 hours after the end of it. Furthermore, the perception of pain and recovery of the lower limbs were also collected at specific moments by means respectively of the Likert scale of perceived effort and visual analogue scale pain. Appropriate statistical analysis was used to compare the groups and the moments, considering the 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Healthy
* Aged between 18 and 30 years
* Classified as physically active through the International Physical Activity Questionnaire

Exclusion Criteria:

* Anemia
* Inflammation
* Diabetes
* Cardiovascular disease
* Liver problems
* Alcoholics
* Smokers
* Illicit drug users
* Chronic users of anti-inflammatory drugs
* Episode of musculotendinous or osteoarticular injury in the lower and/or column members during the last six months.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Creatine kinase using 5 ml samples of blood at 96 hours | 24, 48, 72 and 96 hours after exercise protocol
Change from Baseline in Lactate by means of 25 μl of arterial blood from the ear lobe at 74 minutes | 3, 5, 7, 9, 11, 13, 15, 30, 45, 60 and 75 minutes of achievement of recuperative technique

SECONDARY OUTCOMES:
Change from Baseline in leg pain using the Visual Analogue Scale at 96 hours | 24, 48, 72 and 96 hours after exercise protocol
Change from Baseline in Perception recovery through the scale of perceived effort Likert at 96 hours | 75 minutes, 24, 48, 72 and 96 hours after exercise protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil